CLINICAL TRIAL: NCT04984655
Title: Pilot Study: Virtual Reality Experience for Stress Reduction in Cardiology Patients
Brief Title: Virtual Reality Experience for Stress Reduction in Cardiology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tamara Horwich, Health Sciences Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-000705
Record Dates: First submitted 2021-06-14; First posted 2021-07-30 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Stress; Blood Pressure; Virtual Reality; Prevention

STUDY DESIGN:
Intervention Model Description: Pilot Study (uncontrolled)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30-minute Virtual Reality (VR) Experience delivered through Oculus Quest 2 VR headset (Other)
  Interventions: Device: 30-minute Virtual Reality (VR) Experience delivered through Oculus Quest 2 VR headset

INTERVENTIONS:
Device: 30-minute Virtual Reality (VR) Experience delivered through Oculus Quest 2 VR headset — All participants will go through the same intervention described above

SUMMARY:
The purpose of the research is to evaluate the feasibility and scalability of delivering a 30-minute novel virtual reality (VR) experience through the Oculus Quest 2 Virtual Reality headset with the aim of measuring changes in: 1) patient-reported stress levels on a survey, 2) blood pressure, 3)heart rate, 4) respiration rate 5) heart rate variability 6) and galvanic skin response in cardiology clinic and cardiac rehabilitation patients.

DETAILED DESCRIPTION:
After consenting to participate, participants will be asked to complete a pre-experience questionnaire. The investigators will ask participants questions to evaluate their general and current state of stress as well as gather some baseline health information. Although the questionnaires ask questions about anxiety, they are being conducted for research purposes, so if participants are feeling anxious they should discuss this with their primary care provider or other doctor. The investigators think it should take about 5 minutes to complete the pre-experience questionnaire. If participants feel uncomfortable or embarrassed answering any question, they may skip it. The questionnaire will not contain any information that could be used to identify participants. If participants do not feel comfortable answering surveys then this would result in withdrawal from the study. Participants would be politely notified of your withdrawal and not complete the study.

Participants will then place the VR headset over their head along with over the ear headphones. The research member will ensure safety and comfort then instruct participant how to begin the experience through the headset. The experience includes relaxing images, shapes, and colors that change and evolve slowly. These visuals are also paired with music, which can be adjusted at the start of the experience with the assistance of the researcher (participant will not have to control sound or light). Participants will not have a choice as to the content viewed during this experience. If at any time during the experience participant would like to stop, you may feel free to signal to the researcher, ask to stop, or just remove the headset and headphones.

After completion of the experience, participants will be asked to complete a post-experience survey. Investigators think this should take about 5 minutes to complete. Investigators will again ask about stress levels. Investigators will also gather feedback from participant about thoughts and attitudes towards the VR experience for stress reduction and potential usefulness in cardiac rehabilitation.

Physiological measures will be collected and monitored as follows: The heart rate and heart rate variability will be monitored via the PolarH10 heart rate monitor and chest strap and transmitted to the safely encrypted computer/tablet. There will be no info transmitted with the data aside from the time/date of the collecting. This will be a continuous recording from 5 minutes after you sit down to complete the survey until 5 minutes after the experience. The blood pressure cuff will be used 3 times: 5 minutes after you sit down but prior to the experience, at 15 minutes during the experience, and at the end of the experience. Respiratory rate will be observed by the researcher while you enter the survey data, and every 10 minutes during the experience, then as you complete the post-survey for a total of 5 measurements. The galvanic skin response (sweat gland activity) sensor will be placed at the same time as the heart rate monitor and will provide continuous monitoring for 5 minutes prior to the start of the experience and 5 minutes post-experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current patient in University of California, Los Angeles (UCLA) Cardiology clinics and/or cardiac rehab
* English speaking
* Able to give informed consent

Exclusion Criteria:

* history of seizure
* facial injury preventing safe placement of headset, significant visual or hearing impairment (as defined as not able to see/hear clearly even with corrective lenses/aids).
* Individuals with dangerous, unstable arrhythmias (VTACH/VFIB) and/or myocardial infarction (MI) in past 4 week, or individuals in acute decompensated heart failure
* respiratory issues, postural instability, and motion sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
change in patient-reported stress levels on a survey | immediately before 30-minute virtual reality experience and immediately after 30-minute virtual reality experience

SECONDARY OUTCOMES:
change in systolic blood pressure | immediately before 30-minute virtual reality experience and immediately after 30-minute virtual reality experience
change in diastolic blood pressure | immediately before 30-minute virtual reality experience and immediately after 30-minute virtual reality experience
change in heart rate | immediately before 30-minute virtual reality experience, during the 30-minute virtual reality experience, immediately after 30-minute virtual reality experience
change in heart rate variability | immediately before 30-minute virtual reality experience, during the 30-minute virtual reality experience, immediately after 30-minute virtual reality experience
change in respiration rate | immediately before 30-minute virtual reality experience and immediately after 30-minute virtual reality experience
change in galvanic skin response | immediately before 30-minute virtual reality experience, during the 30-immediately after 30-minute virtual reality experience

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Horwich, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Clinical and Translational Research Center, 10833 Le Conte suite BE144 - CHS building, Los Angeles, California, United States